CLINICAL TRIAL: NCT00951899
Title: The Effect of Colesevelam Hydrochloride on Disposition Index and Incretin Concentrations in Subjects With Type 2 Diabetes Using a Double-blind, Placebo-controlled, Parallel-group Study Design
Brief Title: The Effect of Welchol on Glucose Metabolism in Type 2 Diabetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Daiichi Sankyo (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Adrian Vella, MD, Professor of Medicine, Endocrinology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 08-008284; R01DK078646 (NIH); R01DK082396 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
Keywords: Incretins; colesevelam; hepatobiliary circulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Colesevelam Hydrochloride; Diet; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colesevelam (Experimental): Treatment with colesevelam hydrochloride in addition to Metformin and Diet
  Interventions: Drug: Colesevelam; Behavioral: Diet; Drug: Metformin
- Placebo (Placebo Comparator): Treatment with placebo in addition to Metformin and Diet
  Interventions: Other: Placebo; Behavioral: Diet; Drug: Metformin

INTERVENTIONS:
Drug: Colesevelam — Colesevelam hydrochloride; three 625mg tablets taken orally twice per day before breakfast and before the evening meal over a 12-week treatment period.
  Other Names: Welchol
  Arms: Colesevelam
Other: Placebo — Three placebo tablets matching the active drug colesevelam in appearance, taken orally twice per day before breakfast and before the evening meal over a 12-week treatment period.
  Arms: Placebo
Behavioral: Diet — Subjects were instructed to follow a weight maintenance diet (~55% carbohydrate, 30% fat and 15% protein) for the 12 week study period.
Drug: Metformin — Subjects continued to take their pre-study therapeutic doses of metformin (Metformin 500mg tablets taken by mouth twice daily for a total daily dose of 1000 to 2000 mg) through the 12 week study period.
  Other Names: Glucophage; Glucophage XR; Glumetza; Fortamet

SUMMARY:
The goal of this study was to determine the metabolic mechanism for a certain type medication's ability to lower blood sugar after a meal in Type 2 Diabetics, in order to develop a better understanding of it's potential role in the treatment of obesity.

DETAILED DESCRIPTION:
Welchol (colesevelam hydrochloride) is a bile acid sequestrant (BAS) recently approved by the FDA for glucose lowering in patients with type 2 diabetes mellitus. Four randomized, controlled clinical studies in subjects with type 2 diabetes have demonstrated significant treatment difference in HbA1c (-0.5%). Study durations ranged from 12-26 weeks of therapy. In diabetes clinical studies, a therapeutic response to colesevelam hydrochloride, as reflected by reduction in A1c was initially noted following 4-6 weeks of treatment and reached maximal or near-maximal effect after 12-18 weeks of treatment. Reductions in both fasting plasma glucose and postprandial concentrations have been demonstrated. Simple measures of insulin secretion and action have suggested that this is due to improved insulin action rather than improved insulin secretion. The mechanism by which bile acids interact with the key pathways regulating glucose concentrations is largely unknown. The investigators propose a randomized, double-blind, placebo controlled trial with a parallel-group design where subjects are randomized to receive colesevelam or matching placebo for a 12 week treatment period. A labeled mixed meal before and after treatment will be used to measure intestinal transit, postprandial and fasting glucose fluxes, insulin secretion and action as well as enteroendocrine secretion.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-70 years old.
* Body Mass Index greater than 19kg/m^2 or less than 40kg/m^2 or a total weight less than 130 kilograms.
* Negative pregnancy test for women of childbearing potential.
* Absence of gastrointestinal symptoms.
* Signed informed consent.
* Treatment with diet and/or metformin. Subjects must be on stable therapeutic doses of metformin and/or lipid-lowering agents for more than 3 months.

Exclusion Criteria:

* Structural or metabolic diseases/conditions that affect the gastrointestinal system, or functional gastrointestinal disorders. A screening Bowel Disease Questionnaire will be used to exclude subjects with irritable bowel syndrome. Patients with a history of dysphagia or intestinal motility disorders will be excluded.
* Prior history of pancreatitis.
* Prior history of hypertriglyceridemia (500mg/dL or greater).
* Currently using a bile-acid binding resin such as colesevelam, colestipol, colestimide or cholestyramine.
* To ensure homogeneity between treatment groups we will exclude subjects with insulin-treated type 2 diabetes mellitus, subjects who have received an inhibitors of dipeptidyl peptidase 4 (DPP-4 inhibitors) or "gliptins" (a class of oral hypoglycemics), Byetta or sulfonylurea agent in the past three months.
* HbA1c greater than 9.0%.
* Patients who have not been stable on all medications for a period exceeding 3 months.
* Use of drugs or agents within the past 2 weeks or planned use in the subsequent 4 weeks during the study period that:

  * Alter GI transit including laxatives, magnesium or aluminum-containing antacids, prokinetics, erythromycin, narcotics, anticholinergics, tricyclic antidepressants, Selective Serotonin Reuptake Inhibitors (SSRIs) and newer antidepressants.
  * Opiate-based analgesic drugs (Note: intermittent or chronic use of aspirin or non-steroidal anti-inflammatory drugs (NSAID) will be allowed).
  * Antihistamines
  * Anticholinergic agents
* Female subjects who are pregnant or breast-feeding. Females must be either surgically sterilized, postmenopausal (>12 months since last menses), or, if of childbearing potential, using reliable methods of contraception as determined by the physician.
* Clinical evidence (including physical exam and Electrocardiogram) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric, or other disease that interfere with the objectives of the study. Any candidate participants with such disorders mentioned will be referred to their general physician.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Smushkin G, Sathananthan M, Piccinini F, Dalla Man C, Law JH, Cobelli C, Zinsmeister AR, Rizza RA, Vella A. The effect of a bile acid sequestrant on glucose metabolism in subjects with type 2 diabetes. Diabetes. 2013 Apr;62(4):1094-101. doi: 10.2337/db12-0923. Epub 2012 Dec 18. PMID 23250357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with type 2 diabetes on monotherapy with Metformin were recruited by advertisement from 2009 to 2010 at Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: 39 subjects provided written informed consent to participate. One subject lost intravenous access during the baseline study and withdrew consent. The remaining 38 were randomized.
Groups:
- Colesevelam: Treatment with colesevelam in addition to metformin and diet
- Placebo: Placebo plus diet and metformin
Period: Overall Study
Arm/Group | Colesevelam | Placebo
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for only the randomized subjects (19/19).
Groups:
- Total: Total of all reporting groups
Arm/Group | Colesevelam | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 38
Age Continuous [Mean (Standard Deviation); unit: years] — Age is reported for the randomized subjects only.
  years | 62.6 (5.9) | 60.2 (6.3) | 61 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender reported for only the randomized subjects.
  Participants
    Female | 6 | 6 | 12
    Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is a health index for comparing weight to height. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared. The body mass index is an indication if a person is at a suitable weight for his height on an approximation of body fat.
  kg/m^2 | 30.8 (4.3) | 30.4 (4.0) | 30.6 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Total Disposition Index
Description: Total Disposition Index (DI) is a calculated value which represents the ability of a person's pancreas to lower blood glucose. A higher number means the pancreas is better able to lower blood glucose and a lower number means the pancreas is less able to lower blood glucose.
Time Frame: Baseline, 12 weeks
Population: Intent to treat analysis population.
Measure: Mean (Standard Error); unit: DItot (10^-14 dl/kg/min^2 per pmol/l)
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 19 | 19
DItot (10^-14 dl/kg/min^2 per pmol/l)
  Disposition Index at Baseline | 332 (41) | 253 (40)
  Disposition Index at 12 Weeks | 519 (169) | 310 (48)

2. Secondary Outcome: Total Fasting Glucagon-Like Peptide-1 (GLP-1) Concentration
Description: GLP-1 is thought to increase insulin secretion and was measured in the blood and reported in picomoles per liter.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 19 | 19
pmol/L
  Total GLP-1 at Baseline | 18.3 (1.8) | 18.6 (1.7)
  Total GLP-1 at 12 Weeks | 21.9 (2.1) | 19.3 (2.4)
Statistical Analysis 1: Comparison: Colesevelam; Comparison of mean total GLP-1 concentration from baseline to 12 weeks in Colesevelam subjects; Test type: Superiority or Other; p = 0.0006, t-test, 2 sided — A P value < 0.05 was considered statistically significant
Statistical Analysis 2: Comparison: Placebo; Comparison of mean total GLP-1 concentration from baseline to 12 weeks in Placebo subjects; Test type: Superiority or Other; p = 0.30, t-test, 2 sided

3. Secondary Outcome: Plasma Glucose Concentration
Description: Fasting glucose concentrations were measured at baseline and 2 hours post-meal using the glucose oxidase method.
Time Frame: Baseline, 12 Weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 19 | 19
mmol/L
  Glucose at Baseline | 7.0 (0.2) | 7.4 (0.3)
  Glucose at 12 Weeks | 6.6 (0.2) | 7.5 (0.5)
  Postmeal Glucose Peak at Baseline | 15.4 (0.6) | 15.4 (0.6)
  Postmeal Glucose Peak at 12 Weeks | 14.4 (0.6) | 15.8 (0.6)

4. Secondary Outcome: Glycosylated Hemoglobin (HbA1c)
Description: HbA1c is the percent of red blood cell hemoglobin with glucose attached to it and an indicator of average blood glucose over the previous two to three months.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: Percentage of hemoglobin
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 19 | 19
Percentage of hemoglobin
  HbA1c at Baseline | 6.7 (0.1) | 6.8 (0.1)
  HbA1c at 12 Weeks | 6.5 (0.2) | 6.9 (0.2)

5. Secondary Outcome: Insulin Concentration
Description: Fasting insulin levels were measured in the plasma using a chemiluminescence assay and is reported in nanomoles over 6 hours.
Time Frame: Baseline, 12 Weeks
Measure: Mean (Standard Error); unit: nmols/6 hrs
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 19 | 19
nmols/6 hrs
  Insulin at Baseline | 48 (6) | 50 (6)
  Insulin at 12 Weeks | 45 (5) | 51 (6)
  Postmeal Insulin at Baseline | 67.3 (7.9) | 72.7 (8.3)
  Postmeal Insulin at 12 Weeks | 63.9 (6.1) | 81.9 (11.6)

6. Secondary Outcome: Fasting Endogenous Glucose Production (EGP)
Description: EGP was measured using a triple-tracer mixed meal and calculated using the Steele's model, reported in micromoles per kilogram per minute.
Time Frame: Baseline, 12 Weeks
Measure: Mean (Standard Error); unit: micromol/kg/min
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 19 | 19
micromol/kg/min
  EGP at Baseline | 17.6 (0.6) | 17.7 (0.7)
  EGP at 12 Weeks | 17.2 (0.6) | 17.6 (0.7)

7. Secondary Outcome: Rate of Meal Glucose Appearance (Meal Ra)
Description: Meal Ra was measured using a triple-tracer mixed meal and reported in micromols in 6 hours. Meal derived glucose is a function of both gastric emptying and splanchnic meal extraction. Meal Ra was calculated by multiplying rate of appearance of [1-^13C] glucose (obtained from the infusion rate of [6-^3H] glucose and the clamped plasma ratio of [6-^3H] glucose and [1-^13C] glucose) by the meal enrichment.
Time Frame: Baseline, 12 Weeks
Measure: Mean (Standard Error); unit: micromol/6h
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 19 | 19
micromol/6h
  Meal appearance glucose at Baseline | 5941 (402) | 5504 (354)
  Meal appearance glucose at 12 Weeks | 5413 (289) | 5613 (354)

8. Secondary Outcome: Rate of Meal Glucose Disappearance (Meal Rd)
Description: Meal Rd is the rate at which glucose leaves the systemic circulation. It was measured using a triple-tracer mixed meal and reported in micromols over 6 hours. Meal Rd was calculated by subtracting the change in glucose mass from the overall rate of glucose appearance (i.e., meal Ra + EGP).
Time Frame: Baseline, 12 Weeks
Measure: Mean (Standard Error); unit: micromol/6h
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 19 | 19
micromol/6h
  Meal Rd at Baseline | 8642 (414) | 8784 (403)
  Meal Rd at 12 Weeks | 8155 (314) | 8761 (382)

9. Secondary Outcome: Lipid Values
Description: Lipids are fat-like substances in the blood.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: mmol/l
Arm/Group | Colesevelam | Placebo
Number analyzed (Participants) | 19 | 19
mmol/l
  Total Cholesterol at Baseline | 4.35 (0.19) | 4.33 (0.14)
  Total Cholesterol at 12 weeks | 3.60 (0.16) | 4.00 (0.14)
  Triglycerides at Baseline | 1.67 (0.15) | 1.88 (0.27)
  Triglycerides at 12 Weeks | 2.19 (0.19) | 1.55 (0.18)
  High Density Lipoprotein (HDL) at Baseline | 1.18 (0.06) | 1.27 (0.08)
  High Density Lipoprotein (HDL) at 12 Weeks | 1.08 (0.10) | 1.20 (0.07)
  Low Density Lipoprotein (LDL) at Baseline | 2.50 (0.17) | 2.31 (0.13)
  Low Density Lipoprotein (LDL) at 12 Weeks | 1.59 (0.14) | 2.09 (0.12)

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks.
Arm/Group | Colesevelam | Placebo
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colesevelam (N=19) | Placebo (N=19)
GI ulcer and hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject experienced gastric (antral) ulcerations of unknown etiology, causing melena with acute GI blood loss.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colesevelam (N=19) | Placebo (N=19)
Low hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Low hemoglobin found during visit with primary MD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No